CLINICAL TRIAL: NCT06873399
Title: Machine Learning Assisted Prediction of Keratoconus Progression Using Topographic and Volumetric Data: a Retrospective Study
Brief Title: Detection of Keratoconus Progression Using Machine Learning
Status: Active, not recruiting | Type: Observational
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Head of Department, Vienna Institute for Research in Ocular Surgery
Other Study IDs: EK_24_158_VK
Record Dates: First submitted 2025-03-02; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Keratoconus; Machine Learning
Keywords: keratoconus; machine learning
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Progressive Keratoconus: Patients with progressive keratokonus, based on a one-year change in Kmax values
  Interventions: Diagnostic Test: MS-39
- Non-progressive Keratoconus: Patients with non-progressive keratokonus, based on a one-year change in Kmax values
  Interventions: Diagnostic Test: MS-39

INTERVENTIONS:
Diagnostic Test: MS-39 — The MS-39 (Costruzione Strumenti Oftalmici, Firenze, Italy) is a device for anterior segment analysis of the eye, which combines Placido disc corneal topography and high-resolution SD-OCT. The device provides information on pachymetry, elevation, curvature, and dioptric power of both corneal surfaces. To obtain corneal topography, 22 Placido disc rings are emanated from a laser emitted diode (LED) light source at 635 nanometres (nm). The central 10 millimetres of the anterior corneal surface are covered. Epithelial thickness maps are calculated for different sectors (central, paracentral inferior/superior/nasal/temporal).

SUMMARY:
Keratoconus (KC) is a bilateral ocular disease characterized by progressive thinning and steepening of the cornea, usually in its inferotemporal region. The disease often occurs asymmetrically as one eye is more severely affected by the condition. The changes underlying KC lead to the generation of irregular astigmatism resulting in diminished visual acuity of the patients and can even lead to axial corneal scarring in advanced stages. The disease usually occurs in the second or third decade of life, but can develop at any age. KC is a complex condition involving environmental factors such as age, eye rubbing, contact lens use, atopy, sun exposure, hormones, toxins, as well as a genetic component. However, how these factors contribute to the disease is still unknown and intraindividual differences might exist.

KC can be categorized into different forms based on the stage of the disease. In clinical KC, there are both topographic and slit lamp findings of the disease.

The importance of corneal epithelial imaging in the diagnosis of keratoconus has been further demonstrated in several clinical studies. As new anterior segment optical coherence tomography (AS-OCT) devices provide more detailed measurements for instance of the corneal epithelium. This layer could therefore be an interesting marker for the prediction of KC progression and contribute to earlier diagnosis as well as better outcome of the disease.

The aim of this retrospective study is therefore to determine whether different topographical and volumetric data, for instance epithelial thickness maps (ETM), can be reliably used to predict the progression of KC using a machine learning algorithm.

ELIGIBILITY:
Inclusion Criteria:

* Patients with KC progression as defined dependent on Kmax/year:

o

1. Kmax < 48 Dioptres (D): >0.5 D per year o
2. Kmax 48.01-53 D: >0.6 D per year o
3. Kmax 53.01-58 D: >0.8 D per year o
4. Kmax > 58 D: >1.5 D per year - Non progressive group: Patients with stable KC (KC progression dependent on Kmax < than the values described above/year)

Exclusion Criteria:

* Relevant other ophthalmic diseases that are likely to influence the measurement outcome like corneal scars or epithelial dystrophies
* Too few measurements/too short follow-up to define progression of KC

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with keratoconus that had at least two measurement using the MS-39 device
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of the machine learning algorithm on the final test data set | through study completion, one year
  Sensitivity of the machine learning algorithm on the final test data set to differentiate between progressive/non-progressive eyes based on Kmax-change per year
Specificity of the machine learning algorithm on the final test data set | through study completion, one year
  Specificity of the machine learning algorithm on the final test data set to differentiate between progressive/non-progressive eyes based on Kmax-change per year

CONTACTS AND LOCATIONS:
Locations (1):
- Vienna Institute for Research in Ocular Surgery (VIROS), Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided